CLINICAL TRIAL: NCT01391871
Title: A Randomized Prospective Multicenter Trial to Compare Vascular Healing and Vasodilation at 3 Months After Deployment of PRO-Kinetic Drug-eluting Stent and Endeavor Resolute Zotarolimus-eluting Stent in Patients With Acute Coronary Syndromes by Means of Optical Coherence Tomography and Coronary Flow Reserve
Brief Title: Vascular Healing of DES at 3 Months
Acronym: HAT-TRICK-OCT
Status: Completed | Type: Observational
Sponsor: University of Turku (Other)
Collaborators: The Hospital District of Satakunta (Other)
Responsible Party: Principal Investigator, Tuomas Kiviniemi, MD, PhD, University of Turku
Other Study IDs: HAT-TRICK-OCT
Record Dates: First submitted 2011-07-07; First posted 2011-07-12 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-08

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PRO-Kinetic DES: Patients receiving PRO-Kinetic drug-eluting stent
  Interventions: Device: OCT; Device: Transthoracic echocardiography CFR measurement
- Endeavor Resolute DES: Patient receiving Endeavor Resolute zotarolimus-eluting stent
  Interventions: Device: OCT; Device: Transthoracic echocardiography CFR measurement

INTERVENTIONS:
Device: OCT — Optical coherence tomography
Device: Transthoracic echocardiography CFR measurement — CFR will be assessed using transthoracic echocardiography with adenosine infusion.

SUMMARY:
The purpose of this study is to compare vascular healing of the stented segment after deployment of new PRO-Kinetic drug eluting stent and Endeavor Resolute zotarolimus-eluting stent in patients with acute coronary syndromes requiring percutaneous coronary intervention.

DETAILED DESCRIPTION:
Objective: The aim of the trial is to compare vascular healing and vasodilation at 3 months after deployment of PRO-Kinetic drug-eluting stent and Endeavor Resolute zotarolimus-eluting stent in patients with acute coronary syndrome.

Design: A prospective, randomized and controlled study comparing coronary flow reserve and coverage of the PRO-Kinetic DES and Endeavor Resolute DES implanted in acute coronary syndrome. OCT and CFR measurement at 3 months. Clinical follow up is scheduled at 3, 6 and 12 months.

Primary endpoint: Uncovered stent struts and CFR at 3 months after stent implantation.

Secondary clinical endpoints: MACE and stent thrombosis.

Enrollment: 40 patients (20 receiving PRO-Kinetic DES and 20 receiving Endeavor Resolute DES).

ELIGIBILITY:
Inclusion Criteria:

* STEMI or NSTEMI or unstable angina
* Patient or legally authorized representative has been informed of the nature of the study, agrees to its provisions and has been provided written informed consent, approved by the appropriate Medical Ethics committee or Institutional Review Board.
* Single de novo or non-stented restenosis lesion of LAD
* Patients with two-vessel disease may have undergone successful treatment of the non-target vessel with approved devices up to and including the index procedure but must be treated prior to the index target vessel treatment.
* Target lesion (maximum 20 mm length by visual estimate) to be covered by a single stent of maximum 23mm length.
* Reference vessel diameter must be >2.5mm and <4.0mm by visual estimate.
* The vessel diameter should be measured after pre-dilation procedure and after intracoronary nitroglycerin if vasospasm is suspected.
* Target lesion >50% and <100% stenosed by visual estimate.

Exclusion Criteria:

* Pre-existing diagnosis of diabetes irrespective of its type.
* Impaired renal function (serum creatinine >177micromol/l) or on dialysis
* Platelet count < 10 e5 cells/mm3
* Patient has a history of bleeding diathesis or coagulopathy or patients in whom antiplatelet and and/or anticoagulation therapy is contraindicated.
* Patient has received organ transplant or is on a waiting list for any organ transplant.
* Patient has a known hypersensitivity or contraindication to aspirin, heparin/bivalirudin, clopidogrel/prasugrel, stainless steel alloy, or contrast agent that cannot be adequately pre-medicated.
* Patient presents with cardiogenic shock.
* Any significant medical condition which in the Investigator's opinion may interfere with the patient's optimal participation in the study.
* Currently participating in another investigational drug or device study.
* Unprotected left main disease.
* Ostial target lesions.
* Chronic total occlusion.
* Calcified target lesions that cannot be adequately pre-dilated.
* Target lesion has excessive tortuosity unsuitable for stent delivery and deployment.
* Target lesion involving bifurcation with a side branch larger than 2.0mm in diameter.
* A >30% stenosis proximal or distal to the target lesion that cannot be covered with the same stent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute coronary syndrome treated with PRO-Kinetic DES or Endeavor Resolute DES during index PCI.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2011-06; Primary Completion 2012-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Uncovered stent struts | 3 months
  Percentage of uncovered stent struts per stent by OCT
Coronary flow reserve | 3 months
  Coronary flow reserve by transthoracic echocardiography.

SECONDARY OUTCOMES:
MACE and target vessel stent thrombosis | 12 months
  Death, MI (Q wave or non-Q wave), emergent CABG, or justified TLR by repeat PCI or CABG, and target vessel stent thrombosis.

CONTACTS AND LOCATIONS:
Overall Officials: Tuomas Kiviniemi, MD, PhD, Principal Investigator — Turku University Hospital; Pasi Karjalainen, MD, PhD, Principal Investigator — Satakunta Central Hospital; Antti Ylitalo, MD, PhD, Principal Investigator — Satakunta Central Hospital; Juhani Airaksinen, MD, PhD, FESC, Principal Investigator — Turku University Hospital
Locations (2):
- Finland (2):
  - Satakunta Central Hospital, Pori, Pori
  - Turku University Hospital, Turku